CLINICAL TRIAL: NCT04725006
Title: Sensory Responses to Dorsal Root Stimulation
Status: Withdrawn | Type: Observational
Why Stopped: No participant/patient opportunities for testing. Received funding for a different study.
Sponsor: Lee Fisher, PhD (Other)
Responsible Party: Sponsor-Investigator, Lee Fisher, PhD, Assistant Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Other Study IDs: STUDY20020043
Record Dates: First submitted 2021-01-21; First posted 2021-01-26 (Actual); Last update posted 2025-10-15 (Actual); Status verified 2025-10

CONDITIONS: Amputation; Sensation, Phantom
Keywords: spinal cord stimulation; dorsal root ganglia stimulation; sensation; amputation; pain
MeSH Terms: conditions — Phantom Limb; Pain

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Stimulation in individuals with implanted stimulation systems: During psychophysical stimulation trials, an external stimulator will be connected to the SCS lead, a volley of stimulation will be performed, and the subject will be asked to respond to standard psychophysical questions, as well as to provide any additional comments.
  Interventions: Device: Spinal cord stimulation system

INTERVENTIONS:
Device: Spinal cord stimulation system — These systems are indicated as an aid in the management of chronic intractable pain of the trunk and/or limbs, including unilateral or bilateral pain associated with the following: failed back surgery syndrome, intractable low back pain and leg pain. Stimulation will be applied to the system using an external stimulator to see if sensations can be evoked in the participant's limb/foot.
  Other Names: Boston Scientific; St. Jude

SUMMARY:
The goal of this project is to characterize the types of sensations that can be evoked via electrical stimulation of the spinal cord and spinal nerves. Patients will be recruited from a local pain clinic, each with a spinal cord stimulation device implanted, to participate in experiments to explore the ability to modulate and control the modality, intensity, focality, and location of the sensations evoked by stimulation through the spinal cord stimulator leads. Investigators will connect spinal cord stimulator leads to a custom stimulator system and will ask subjects to report the types of sensations felt. Invesigators will also perform detailed psychophysical metrics to examine participants' ability to discriminate sensations.

DETAILED DESCRIPTION:
For this study, investigators aim to determine whether DRG and spinal root stimulation might be viable techniques for restoring feedback. Investigators will focus on patients undergoing temporary percutaneous trials of DRG or lateral spinal cord stimulation with leads manufactured by either Boston Scientific (under PMA P030017) or St. Jude (under PMA P150004), which have FDA premarket approval for the management of chronic pain in the trunk and lower limbs. In this early experiment, investigators will not focus on individuals with limb loss, but rather will include patients already undergoing a percutaneous trial of DRG or spinal root stimulation to treat pain. Investigators will characterize the location, modality, and intensity of sensations evoked in the hands or feet with stimulation delivered by an external stimulator.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must be between the ages of 18 and 70 years old.
2. Subjects must be undergoing an epidural spinal cord implanted electrode array clinical trial with Dr. Helm for the management of pain.
3. Persons must understand the consent and the procedures.

Exclusion Criteria:

1. Persons with open wounds;
2. Persons with implanted metal rods in the spine or limbs;
3. Persons with defibrillator or pacemaker;
4. Persons with permanent skin metal tags or decorations.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals undergoing a 7-day trial period of percutaneous DRG or spinal root stimulation.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2020-12-16 (Actual); Primary Completion 2025-07-11 (Actual); Study Completion 2025-10-07 (Actual)

PRIMARY OUTCOMES:
Location of evoked sensory percepts | up to 2 days
  Document where on the body the subject perceives the stimulation locations.
Stimulation perceptual thresholds to stimulus parameters | up to 2 days
  Quantify the threshold stimulus required to evoke sensory percepts during epidural spinal nerve stimulation.
Stimulation neurophysiology thresholds to stimulus parameters | up to 2 days
  Quantify the threshold stimulus required to evoke neurophysiological responses during epidural spinal nerve stimulation

SECONDARY OUTCOMES:
Qualitative self-report of evoked sensations | up to 2 days
  Document the subjective perception of lumbosacral epidural spinal nerve stimulation for restoration of sensation. The investigators will ask each subject to provide subjective feedback on their perceived utility of the sensory feedback provided by the device.

CONTACTS AND LOCATIONS:
Overall Officials: Lee Fisher, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No